CLINICAL TRIAL: NCT05618626
Title: Cardiovascular Diseases (CVD) and Nonalcoholic Fatty Liver Diseases (NAFLD) Among Gallstone and Cholecystectomy Patients and the Impact of a Novel Diet and Muscle Training Program
Brief Title: Prevention of NAFLD and CVD Through Lifestyle Intervention
Acronym: MAUCO+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Catterina Ferreccio, Principal Investigator, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FN1212066
Record Dates: First submitted 2022-06-17; First posted 2022-11-16 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Gallstone Disease
Keywords: Anti-inflammatory diet; Lifestyle modification; Physical Activity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Cholelithiasis; Motor Activity | interventions — Exercise; Diet Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical exercise and dietary intervention for NAFLD (Experimental): The exercise program will consist of muscular strength and aerobic exercises; additionally, each session will start and end with low intensity warm-up and cool down periods. The program will be divided in months. Months 1-2, twice a week directly-supervised exercises group sessions, and 1 telehealth session. Months 3-6, once a week directly-supervised group session and twice a week home-based telehealth. Months 7-12, Monthly telephone support. Months 12, 24 and 36, All participants (control and intervention arms) will receive a full evaluation. In the dietary intervention, investigators proposed a diet rich in anti-inflammatory components, legumes and in dietary fiber. The baseline evaluation of nutritional condition includes: anthropometry, bioimpedance analysis, hepatobiliary ultrasound, Fibroscan,blood lipids, and a battery of metabolic markers and a diet survey, Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24). Both interventions are performed in parallel.
  Interventions: Other: Physical exercise and dietary intervention for NAFLD
- Standard of care (No Intervention): Participants in the control arm first have a baseline evaluation of the nutritional condition, with anthropometry evaluation, bioimpedance analysis, hepatobiliary ultrasound, Fibroscan, blood lipids, a battery of metabolic markers, and a diet survey, Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24). After the evaluation period, participants received one counseling session, including written material, with advice to follow a healthy diet rich in fruits and vegetables, whole-grain foods, low in salt and sugars, and recommendations for an exercise plan of at least 30 minutes of aerobic exercise three times a week.

INTERVENTIONS:
Other: Physical exercise and dietary intervention for NAFLD — Investigators will assess the efficiency of the intervention by measuring adherence to physical exercise and nutritional diet.
  Arms: Physical exercise and dietary intervention for NAFLD

SUMMARY:
Prevention of non-alcoholic fatty liver disease (NAFLD) and cardiovascular disease (CVD) through lifestyle intervention (MAUCO+) is a clinical trial that aims to improve sarcopenia, aerobic capacity, body composition, and lipid profile, insulin resistance, cardiovascular risk, NAFLD, and maintain a healthier lifestyle. Through the implementation of physical activity and nutritional programs.

DETAILED DESCRIPTION:
BACKGROUND. Gallstone disease (GSD), including gallstones and cholecystectomy, is a common digestive disease worldwide, and Chile has one of the highest reported rates of gallstone prevalence. GSD, in particular cholecystectomy, has been associated with nonalcoholic fatty liver disease (NAFLD). In previous studies, investigators confirmed the association of cholecystectomy with a higher risk of NAFLD only in men. Additionally, reasearchers found a higher cardiovascular event risk in 3 years for male gallstone carriers. Investigators aim to step forward toward translational research by evaluating the effectiveness of a risk-reduction strategy customized to our population.

STUDY GOALS. To evaluate a metabolic risk reduction strategy based on: 1. A Physical exercise trial to increase muscle mass and strength, and 2. A nutritional intervention based on an anti-inflammatory diet, sleep hygiene, and prolonged fasting periods.

METHODS. Intensive Lifestyle Intervention, Randomized Controlled Trial: 300 participants will be randomly allocated to control (n=150) or an experimental group (n=150). The control group will receive standard prevention recommendations, personalized advice, educational material regarding lifestyle and metabolic diseases, and follow-up evaluation of physical activity, physical condition, anthropometry, diet, and sleep habits. The intervention group will receive, tailored to each participant: 3.1 An Exercise Program consisting of directly supervised and home-based telehealth sessions emphasizing muscle building, and 3.2. A Nutritional plus Program based on a diet rich in anti-inflammatory components and legumes, low in fat and refined carbohydrates, controlled energy according to BMI, extended nocturnal fasting periods, and healthy sleep habits. The programs will have a 6-month intensive phase of bi-weekly directly supervised exercise sessions in a municipality gym and a weekly telehealth session, followed by six months of telephone support and bi-monthly direct supervision to reinforce adherence and early identification of risk factors for abandonment. Intervention outcomes measured at baseline and years 1 and 2 are changes in non-invasive serum and ultrasound-based biomarkers of NAFLD; improvement in sarcopenia, aerobic capacity, body composition, lipid profile, insulin resistance, and cardiovascular risk; among overweight participants, permanent loss of at least 5% body weight; the decrease of depression symptoms, improvement of quality of life scores, and maintenance of a healthier lifestyle.

EXPECTED RESULTS: is expected that a 12-month intervention of a personalized physical activity program together with a metabolic protective diet will improve markers of metabolic syndrome and NAFLD and decrease CVD risk scores in all participants who adhere to more than 50% of both interventions, with a clear dose-response effect.

ELIGIBILITY:
Inclusion Criteria:

* With and without gallstones disease
* With various degrees of NAFLD (none too severe)

Exclusion Criteria:

* Any significant comorbidity or physical limitation to undergo resistance exercise program
* Use of medications that alter muscle mass (e.g., corticosteroids)
* History of hepatitis B or C
* Use of hepatotoxic drugs

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Presence and severity of Non-Alcoholic Fatty liver Disease (NAFLD) at baseline and 12 month later. | 36 months
  It will be measured through the liver steatosis marker "Controlled Attenuation Parameter (CAP)" (dB/m).

SECONDARY OUTCOMES:
Framingham Cardiovascular risk score | 36 months
  It will be measured at baseline and 12 months.
HDL cholesterol (mg/dL) | 36 months
  It will be measured at baseline and 12 months.
Triglycerides (mg/dL) | 36 months
  It will be measured at baseline and 12 months.
Glycemia (mg/dL) | 36 months
  It will be measured at baseline and 12 months.
Insulin (uU/mL) | 36 months
  It will be measured at baseline and 12 months.
HBA1c | 36 months
  It will be measured at baseline and 12 months.
usPCR (mg/L) | 36 months
  It will be measured at baseline and 12 months.
AST:ALT ratio | 36 months
  It will be measured at baseline and 12 months.
Total cholesterol (mg/dL) | 36 months
  It will be measured at baseline and 12 months.
Platelets (#cells/uL) | 36 months
  It will be measured at baseline and 12 months.
HOMA-IR | 36 months
  It will be measured at baseline and 12 months.
Total Bilirrubin (mg/dL) | 36 months
  It will be measured at baseline and 12 months.
Alkaline phosphatase (UI/l) | 36 months
  It will be measured at baseline and 12 months.
Glutamiz oxaloacetic transaminase (GOT) (UI/l) | 36 months
  It will be measured at baseline and 12 months.
Glutamic pyruvic trasaminase (GPT) (UI/l) | 36 months
  It will be measured at baseline and 12 months.
Gamma-glutamyl Transferase (GGT) (UI/l) | 36 months
  It will be measured at baseline and 12 months.
Metabolic syndrome | 36 months
  To be diagnosed with metabolic syndrome it is necessary to meet 3 or more conditions. (abdominal obesity, high triglycerides, low HDL cholesterol, high blood pressure and high fasting glucose). Metabolic syndrome will be measure at baseline and 12 month.

OTHER OUTCOMES:
Muscular mass percentage measure | 36 months
  Muscular mass percentage will be measure by bioimpedance analysis at baseline and 12 month.
Body fat percentage | 36 months
  Body fat percentage will be measure by bioimpedance analysis at baseline and 12 month.
Body Mass Index (BMI) (kg/m^2) | 36 months
  A BMI will considered Underweight, Normal, Overweight or Obesity if it is less than 18.5 kg/m^2, it is between 18.5 and 24.9 kg/m^2, it is between 25 and 29.9 kg/m^2, or it is equal or greater than 30 kg/m^2, respectively.
Aerobic capacity VO2max (ml/kg/min) | 36 months
  Aerobic capacity VO2max will be measure at baseline and 12 month
Waist circumference (cm) | 36 months
  Waist circumference will be measure at baseline and 12 month.

CONTACTS AND LOCATIONS:
Overall Officials: Catterina Ferreccio, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Centro MAUCO+, Molina, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stinton LM, Shaffer EA. Epidemiology of gallbladder disease: cholelithiasis and cancer. Gut Liver. 2012 Apr;6(2):172-87. doi: 10.5009/gnl.2012.6.2.172. Epub 2012 Apr 17. PMID 22570746
- [Background] Latorre S G, Ivanovic-Zuvic S D, Corsi S O, Valdivia C G, Margozzini M P, Olea O R, Chianale B J, Miquel P JF. [Coverage of the gallbladder cancer prevention strategy in Chile: results from the 2009-2010 National Health Survey]. Rev Med Chil. 2015 Feb;143(2):158-67. doi: 10.4067/S0034-98872015000200002. Spanish. PMID 25860357
- [Background] Bertran E, Heise K, Andia ME, Ferreccio C. Gallbladder cancer: incidence and survival in a high-risk area of Chile. Int J Cancer. 2010 Nov 15;127(10):2446-54. doi: 10.1002/ijc.25421. PMID 20473911
- [Background] Hundal R, Shaffer EA. Gallbladder cancer: epidemiology and outcome. Clin Epidemiol. 2014 Mar 7;6:99-109. doi: 10.2147/CLEP.S37357. eCollection 2014. PMID 24634588
- [Background] Lammert F, Gurusamy K, Ko CW, Miquel JF, Mendez-Sanchez N, Portincasa P, van Erpecum KJ, van Laarhoven CJ, Wang DQ. Gallstones. Nat Rev Dis Primers. 2016 Apr 28;2:16024. doi: 10.1038/nrdp.2016.24. PMID 27121416
- [Background] Buch S, Schafmayer C, Volzke H, Becker C, Franke A, von Eller-Eberstein H, Kluck C, Bassmann I, Brosch M, Lammert F, Miquel JF, Nervi F, Wittig M, Rosskopf D, Timm B, Holl C, Seeger M, ElSharawy A, Lu T, Egberts J, Fandrich F, Folsch UR, Krawczak M, Schreiber S, Nurnberg P, Tepel J, Hampe J. A genome-wide association scan identifies the hepatic cholesterol transporter ABCG8 as a susceptibility factor for human gallstone disease. Nat Genet. 2007 Aug;39(8):995-9. doi: 10.1038/ng2101. Epub 2007 Jul 15. PMID 17632509
- [Background] Bustos BI, Perez-Palma E, Buch S, Azocar L, Riveras E, Ugarte GD, Toliat M, Nurnberg P, Lieb W, Franke A, Hinz S, Burmeister G, von Schonfels W, Schafmayer C, Volzke H, Volker U, Homuth G, Lerch MM, Santos JL, Puschel K, Bambs C, Roa JC, Gutierrez RA, Hampe J, De Ferrari GV, Miquel JF. Variants in ABCG8 and TRAF3 genes confer risk for gallstone disease in admixed Latinos with Mapuche Native American ancestry. Sci Rep. 2019 Jan 28;9(1):772. doi: 10.1038/s41598-018-35852-z. PMID 30692554
- [Background] Nervi F, Miquel JF, Alvarez M, Ferreccio C, Garcia-Zattera MJ, Gonzalez R, Perez-Ayuso RM, Rigotti A, Villarroel L. Gallbladder disease is associated with insulin resistance in a high risk Hispanic population. J Hepatol. 2006 Aug;45(2):299-305. doi: 10.1016/j.jhep.2006.01.026. Epub 2006 Feb 17. PMID 16516330
- [Background] Lin IC, Yang YW, Wu MF, Yeh YH, Liou JC, Lin YL, Chiang CH. The association of metabolic syndrome and its factors with gallstone disease. BMC Fam Pract. 2014 Jul 29;15:138. doi: 10.1186/1471-2296-15-138. PMID 25070766
- [Background] Shaffer EA. Epidemiology and risk factors for gallstone disease: has the paradigm changed in the 21st century? Curr Gastroenterol Rep. 2005 May;7(2):132-40. doi: 10.1007/s11894-005-0051-8. PMID 15802102
- [Background] Haas JT, Francque S, Staels B. Pathophysiology and Mechanisms of Nonalcoholic Fatty Liver Disease. Annu Rev Physiol. 2016;78:181-205. doi: 10.1146/annurev-physiol-021115-105331. Epub 2015 Nov 30. PMID 26667070
- [Background] Riquelme A, Arrese M, Soza A, Morales A, Baudrand R, Perez-Ayuso RM, Gonzalez R, Alvarez M, Hernandez V, Garcia-Zattera MJ, Otarola F, Medina B, Rigotti A, Miquel JF, Marshall G, Nervi F. Non-alcoholic fatty liver disease and its association with obesity, insulin resistance and increased serum levels of C-reactive protein in Hispanics. Liver Int. 2009 Jan;29(1):82-8. doi: 10.1111/j.1478-3231.2008.01823.x. Epub 2008 Jul 16. PMID 18647235
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] Bellentani S. The epidemiology of non-alcoholic fatty liver disease. Liver Int. 2017 Jan;37 Suppl 1:81-84. doi: 10.1111/liv.13299. PMID 28052624
- [Background] Arrese M, Cortes V, Barrera F, Nervi F. Nonalcoholic fatty liver disease, cholesterol gallstones, and cholecystectomy: new insights on a complex relationship. Curr Opin Gastroenterol. 2018 Mar;34(2):90-96. doi: 10.1097/MOG.0000000000000416. PMID 29266009
- [Background] Brunt EM. Pathology of nonalcoholic fatty liver disease. Nat Rev Gastroenterol Hepatol. 2010 Apr;7(4):195-203. doi: 10.1038/nrgastro.2010.21. Epub 2010 Mar 2. PMID 20195271
- [Background] Koller T, Kollerova J, Hlavaty T, Huorka M, Payer J. Cholelithiasis and markers of nonalcoholic fatty liver disease in patients with metabolic risk factors. Scand J Gastroenterol. 2012 Feb;47(2):197-203. doi: 10.3109/00365521.2011.643481. Epub 2011 Dec 19. PMID 22182015
- [Background] Liu J, Lin H, Zhang C, Wang L, Wu S, Zhang D, Tang F, Xue F, Liu Y. Non-alcoholic fatty liver disease associated with gallstones in females rather than males: a longitudinal cohort study in Chinese urban population. BMC Gastroenterol. 2014 Dec 13;14:213. doi: 10.1186/s12876-014-0213-y. PMID 25496394
- [Background] Chang Y, Noh YH, Suh BS, Kim Y, Sung E, Jung HS, Kim CW, Kwon MJ, Yun KE, Noh JW, Shin H, Cho YK, Ryu S. Bidirectional Association between Nonalcoholic Fatty Liver Disease and Gallstone Disease: A Cohort Study. J Clin Med. 2018 Nov 21;7(11):458. doi: 10.3390/jcm7110458. PMID 30469392
- [Background] Joseph P, Leong D, McKee M, Anand SS, Schwalm JD, Teo K, Mente A, Yusuf S. Reducing the Global Burden of Cardiovascular Disease, Part 1: The Epidemiology and Risk Factors. Circ Res. 2017 Sep 1;121(6):677-694. doi: 10.1161/CIRCRESAHA.117.308903. PMID 28860318
- [Background] Fairfield CJ, Wigmore SJ, Harrison EM. Gallstone Disease and the Risk of Cardiovascular Disease. Sci Rep. 2019 Apr 9;9(1):5830. doi: 10.1038/s41598-019-42327-2. PMID 30967586
- [Background] Lv J, Qi L, Yu C, Guo Y, Bian Z, Chen Y, Yang L, Shen J, Wang S, Li M, Liu Y, Zhang L, Chen J, Chen Z, Li L; China Kadoorie Biobank Collaborative Group*. Gallstone Disease and the Risk of Ischemic Heart Disease. Arterioscler Thromb Vasc Biol. 2015 Oct;35(10):2232-7. doi: 10.1161/ATVBAHA.115.306043. Epub 2015 Aug 13. PMID 26272939
- [Background] Olaiya MT, Chiou HY, Jeng JS, Lien LM, Hsieh FI. Significantly increased risk of cardiovascular disease among patients with gallstone disease: a population-based cohort study. PLoS One. 2013 Oct 3;8(10):e76448. doi: 10.1371/journal.pone.0076448. eCollection 2013. PMID 24098504
- [Background] Shabanzadeh DM, Skaaby T, Sorensen LT, Jorgensen T. Screen-detected gallstone disease and cardiovascular disease. Eur J Epidemiol. 2017 Jun;32(6):501-510. doi: 10.1007/s10654-017-0263-x. Epub 2017 May 27. PMID 28551778
- [Background] Wirth J, di Giuseppe R, Wientzek A, Katzke VA, Kloss M, Kaaks R, Boeing H, Weikert C. Presence of gallstones and the risk of cardiovascular diseases: The EPIC-Germany cohort study. Eur J Prev Cardiol. 2015 Mar;22(3):326-34. doi: 10.1177/2047487313512218. Epub 2013 Oct 31. PMID 24177267
- [Background] Zheng Y, Xu M, Heianza Y, Ma W, Wang T, Sun D, Albert CM, Hu FB, Rexrode KM, Manson JE, Qi L. Gallstone disease and increased risk of mortality: Two large prospective studies in US men and women. J Gastroenterol Hepatol. 2018 Nov;33(11):1925-1931. doi: 10.1111/jgh.14264. Epub 2018 May 27. PMID 29671893
- [Background] Ruhl CE, Everhart JE. Relationship of non-alcoholic fatty liver disease with cholecystectomy in the US population. Am J Gastroenterol. 2013 Jun;108(6):952-8. doi: 10.1038/ajg.2013.70. Epub 2013 Apr 2. PMID 23545713
- [Background] Yue W, Sun X, Du T. Cholecystectomy versus central obesity or insulin resistance in relation to the risk of nonalcoholic fatty liver disease: the third US National Health and Nutrition Examination Survey. BMC Endocr Disord. 2019 Sep 2;19(1):95. doi: 10.1186/s12902-019-0423-y. PMID 31477078
- [Background] Di Ciaula A, Garruti G, Wang DQ, Portincasa P. Cholecystectomy and risk of metabolic syndrome. Eur J Intern Med. 2018 Jul;53:3-11. doi: 10.1016/j.ejim.2018.04.019. Epub 2018 Apr 26. PMID 29706426
- [Background] Nervi F, Arrese M. Cholecystectomy and NAFLD: does gallbladder removal have metabolic consequences? Am J Gastroenterol. 2013 Jun;108(6):959-61. doi: 10.1038/ajg.2013.84. PMID 23735917
- [Background] Barrera F, Azocar L, Molina H, Schalper KA, Ocares M, Liberona J, Villarroel L, Pimentel F, Perez-Ayuso RM, Nervi F, Groen AK, Miquel JF. Effect of cholecystectomy on bile acid synthesis and circulating levels of fibroblast growth factor 19. Ann Hepatol. 2015 Sep-Oct;14(5):710-21. PMID 26256900
- [Background] Ioannou GN. Cholelithiasis, cholecystectomy, and liver disease. Am J Gastroenterol. 2010 Jun;105(6):1364-73. doi: 10.1038/ajg.2009.737. Epub 2010 Jan 12. PMID 20068558
- [Background] Kwak MS, Kim D, Chung GE, Kim W, Kim YJ, Yoon JH. Cholecystectomy is independently associated with nonalcoholic fatty liver disease in an Asian population. World J Gastroenterol. 2015 May 28;21(20):6287-95. doi: 10.3748/wjg.v21.i20.6287. PMID 26034364
- [Background] Cortes V, Quezada N, Uribe S, Arrese M, Nervi F. Effect of cholecystectomy on hepatic fat accumulation and insulin resistance in non-obese Hispanic patients: a pilot study. Lipids Health Dis. 2017 Jun 30;16(1):129. doi: 10.1186/s12944-017-0525-3. PMID 28666456
- [Background] Nishtar S, Niinisto S, Sirisena M, Vazquez T, Skvortsova V, Rubinstein A, Mogae FG, Mattila P, Ghazizadeh Hashemi SH, Kariuki S, Narro Robles J, Adewole IF, Sarr AD, Gan KY, Piukala SM, Al Owais ARBM, Hargan E, Alleyne G, Alwan A, Bernaert A, Bloomberg M, Dain K, Frieden T, Patel VH, Kennedy A, Kickbusch I; Commissioners of the WHO Independent High-Level Commission on NCDs. Time to deliver: report of the WHO Independent High-Level Commission on NCDs. Lancet. 2018 Jul 21;392(10143):245-252. doi: 10.1016/S0140-6736(18)31258-3. Epub 2018 Jun 1. No abstract available. PMID 29866374
- [Background] Brandhorst S, Longo VD. Dietary Restrictions and Nutrition in the Prevention and Treatment of Cardiovascular Disease. Circ Res. 2019 Mar 15;124(6):952-965. doi: 10.1161/CIRCRESAHA.118.313352. PMID 30870119
- [Background] Correction to: 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e649-e650. doi: 10.1161/CIR.0000000000000725. Epub 2019 Sep 9. No abstract available. PMID 31498691
- [Background] Chiuve SE, Fung TT, Rimm EB, Hu FB, McCullough ML, Wang M, Stampfer MJ, Willett WC. Alternative dietary indices both strongly predict risk of chronic disease. J Nutr. 2012 Jun;142(6):1009-18. doi: 10.3945/jn.111.157222. Epub 2012 Apr 18. PMID 22513989
- [Background] Suarez M, Boque N, Del Bas JM, Mayneris-Perxachs J, Arola L, Caimari A. Mediterranean Diet and Multi-Ingredient-Based Interventions for the Management of Non-Alcoholic Fatty Liver Disease. Nutrients. 2017 Sep 22;9(10):1052. doi: 10.3390/nu9101052. PMID 28937599
- [Background] Vilar-Gomez E, Martinez-Perez Y, Calzadilla-Bertot L, Torres-Gonzalez A, Gra-Oramas B, Gonzalez-Fabian L, Friedman SL, Diago M, Romero-Gomez M. Weight Loss Through Lifestyle Modification Significantly Reduces Features of Nonalcoholic Steatohepatitis. Gastroenterology. 2015 Aug;149(2):367-78.e5; quiz e14-5. doi: 10.1053/j.gastro.2015.04.005. Epub 2015 Apr 10. PMID 25865049
- [Background] Tabung FK, Steck SE, Zhang J, Ma Y, Liese AD, Agalliu I, Hingle M, Hou L, Hurley TG, Jiao L, Martin LW, Millen AE, Park HL, Rosal MC, Shikany JM, Shivappa N, Ockene JK, Hebert JR. Construct validation of the dietary inflammatory index among postmenopausal women. Ann Epidemiol. 2015 Jun;25(6):398-405. doi: 10.1016/j.annepidem.2015.03.009. Epub 2015 Mar 19. PMID 25900255
- [Background] Luu HN, Wen W, Li H, Dai Q, Yang G, Cai Q, Xiang YB, Gao YT, Zheng W, Shu XO. Are dietary antioxidant intake indices correlated to oxidative stress and inflammatory marker levels? Antioxid Redox Signal. 2015 Apr 10;22(11):951-9. doi: 10.1089/ars.2014.6212. Epub 2015 Feb 27. PMID 25602689
- [Background] Richard C, Royer MM, Couture P, Cianflone K, Rezvani R, Desroches S, Lamarche B. Effect of the Mediterranean diet on plasma adipokine concentrations in men with metabolic syndrome. Metabolism. 2013 Dec;62(12):1803-10. doi: 10.1016/j.metabol.2013.07.012. Epub 2013 Aug 29. PMID 23993420
- [Background] Casas R, Sacanella E, Estruch R. The immune protective effect of the Mediterranean diet against chronic low-grade inflammatory diseases. Endocr Metab Immune Disord Drug Targets. 2014;14(4):245-54. doi: 10.2174/1871530314666140922153350. PMID 25244229
- [Background] Mirmiran P, Amirhamidi Z, Ejtahed HS, Bahadoran Z, Azizi F. Relationship between Diet and Non-alcoholic Fatty Liver Disease: A Review Article. Iran J Public Health. 2017 Aug;46(8):1007-1017. PMID 28894701
- [Background] Adriano LS, Sampaio HA, Arruda SP, Portela CL, de Melo MLP, Carioca AA, Soares NT. Healthy dietary pattern is inversely associated with non-alcoholic fatty liver disease in elderly. Br J Nutr. 2016 Jun;115(12):2189-95. doi: 10.1017/S0007114516001410. Epub 2016 Apr 22. PMID 27102566
- [Background] Promrat K, Kleiner DE, Niemeier HM, Jackvony E, Kearns M, Wands JR, Fava JL, Wing RR. Randomized controlled trial testing the effects of weight loss on nonalcoholic steatohepatitis. Hepatology. 2010 Jan;51(1):121-9. doi: 10.1002/hep.23276. PMID 19827166
- [Background] Lazo M, Solga SF, Horska A, Bonekamp S, Diehl AM, Brancati FL, Wagenknecht LE, Pi-Sunyer FX, Kahn SE, Clark JM; Fatty Liver Subgroup of the Look AHEAD Research Group. Effect of a 12-month intensive lifestyle intervention on hepatic steatosis in adults with type 2 diabetes. Diabetes Care. 2010 Oct;33(10):2156-63. doi: 10.2337/dc10-0856. Epub 2010 Jul 27. PMID 20664019
- [Background] Perdomo CM, Fruhbeck G, Escalada J. Impact of Nutritional Changes on Nonalcoholic Fatty Liver Disease. Nutrients. 2019 Mar 21;11(3):677. doi: 10.3390/nu11030677. PMID 30901929
- [Background] Bahrami A, Teymoori F, Eslamparast T, Sohrab G, Hejazi E, Poustchi H, Hekmatdoost A. Legume intake and risk of nonalcoholic fatty liver disease. Indian J Gastroenterol. 2019 Feb;38(1):55-60. doi: 10.1007/s12664-019-00937-8. Epub 2019 Feb 22. PMID 30796701
- [Background] Imai S. Soybean and Processed Soy Foods Ingredients, and Their Role in Cardiometabolic Risk Prevention. Recent Pat Food Nutr Agric. 2015;7(2):75-82. doi: 10.2174/2212798407666150629123839. PMID 26118770
- [Background] Ganesan K, Xu B. Polyphenol-Rich Lentils and Their Health Promoting Effects. Int J Mol Sci. 2017 Nov 10;18(11):2390. doi: 10.3390/ijms18112390. PMID 29125587
- [Background] Ganesan K, Xu B. Polyphenol-Rich Dry Common Beans (Phaseolus vulgaris L.) and Their Health Benefits. Int J Mol Sci. 2017 Nov 4;18(11):2331. doi: 10.3390/ijms18112331. PMID 29113066
- [Background] Higgins JA. Resistant starch: metabolic effects and potential health benefits. J AOAC Int. 2004 May-Jun;87(3):761-8. PMID 15287677
- [Background] Martinez I, Kim J, Duffy PR, Schlegel VL, Walter J. Resistant starches types 2 and 4 have differential effects on the composition of the fecal microbiota in human subjects. PLoS One. 2010 Nov 29;5(11):e15046. doi: 10.1371/journal.pone.0015046. PMID 21151493
- [Background] Raghavendra CK, Srinivasan K. Influence of dietary tender cluster beans (Cyamopsis tetragonoloba) on biliary proteins, bile acid synthesis and cholesterol crystal growth in rat bile. Steroids. 2015 Feb;94:21-30. doi: 10.1016/j.steroids.2014.12.003. Epub 2014 Dec 19. PMID 25534812
- [Background] Mvondo MA, Njamen D, Kretzschmar G, Imma Bader M, Tanee Fomum S, Wandji J, Vollmer G. Alpinumisoflavone and abyssinone V 4'-methylether derived from Erythrina lysistemon (Fabaceae) promote HDL-cholesterol synthesis and prevent cholesterol gallstone formation in ovariectomized rats. J Pharm Pharmacol. 2015 Jul;67(7):990-6. doi: 10.1111/jphp.12386. Epub 2015 Feb 14. PMID 25683903
- [Background] Couto Alves A, Glastonbury CA, El-Sayed Moustafa JS, Small KS. Fasting and time of day independently modulate circadian rhythm relevant gene expression in adipose and skin tissue. BMC Genomics. 2018 Sep 7;19(1):659. doi: 10.1186/s12864-018-4997-y. PMID 30193568
- [Background] Marinac CR, Natarajan L, Sears DD, Gallo LC, Hartman SJ, Arredondo E, Patterson RE. Prolonged Nightly Fasting and Breast Cancer Risk: Findings from NHANES (2009-2010). Cancer Epidemiol Biomarkers Prev. 2015 May;24(5):783-9. doi: 10.1158/1055-9965.EPI-14-1292. Epub 2015 Apr 20. PMID 25896523
- [Background] de Cabo R, Mattson MP. Effects of Intermittent Fasting on Health, Aging, and Disease. N Engl J Med. 2019 Dec 26;381(26):2541-2551. doi: 10.1056/NEJMra1905136. No abstract available. PMID 31881139
- [Background] Cai H, Qin YL, Shi ZY, Chen JH, Zeng MJ, Zhou W, Chen RQ, Chen ZY. Effects of alternate-day fasting on body weight and dyslipidaemia in patients with non-alcoholic fatty liver disease: a randomised controlled trial. BMC Gastroenterol. 2019 Dec 18;19(1):219. doi: 10.1186/s12876-019-1132-8. PMID 31852444
- [Background] Alam I, Gul R, Chong J, Tan CTY, Chin HX, Wong G, Doggui R, Larbi A. Recurrent circadian fasting (RCF) improves blood pressure, biomarkers of cardiometabolic risk and regulates inflammation in men. J Transl Med. 2019 Aug 19;17(1):272. doi: 10.1186/s12967-019-2007-z. PMID 31426866
- [Background] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Background] Hutchison AT, Regmi P, Manoogian ENC, Fleischer JG, Wittert GA, Panda S, Heilbronn LK. Time-Restricted Feeding Improves Glucose Tolerance in Men at Risk for Type 2 Diabetes: A Randomized Crossover Trial. Obesity (Silver Spring). 2019 May;27(5):724-732. doi: 10.1002/oby.22449. Epub 2019 Apr 19. PMID 31002478
- [Background] Mazzoccoli G, De Cosmo S, Mazza T. The Biological Clock: A Pivotal Hub in Non-alcoholic Fatty Liver Disease Pathogenesis. Front Physiol. 2018 Mar 15;9:193. doi: 10.3389/fphys.2018.00193. eCollection 2018. PMID 29662454
- [Background] Gnocchi D, Custodero C, Sabba C, Mazzocca A. Circadian rhythms: a possible new player in non-alcoholic fatty liver disease pathophysiology. J Mol Med (Berl). 2019 Jun;97(6):741-759. doi: 10.1007/s00109-019-01780-2. Epub 2019 Apr 5. PMID 30953079
- [Background] Trovato FM, Martines GF, Brischetto D, Trovato G, Catalano D. Neglected features of lifestyle: Their relevance in non-alcoholic fatty liver disease. World J Hepatol. 2016 Nov 28;8(33):1459-1465. doi: 10.4254/wjh.v8.i33.1459. PMID 27957244
- [Background] Hong HC, Hwang SY, Choi HY, Yoo HJ, Seo JA, Kim SG, Kim NH, Baik SH, Choi DS, Choi KM. Relationship between sarcopenia and nonalcoholic fatty liver disease: the Korean Sarcopenic Obesity Study. Hepatology. 2014 May;59(5):1772-8. doi: 10.1002/hep.26716. Epub 2014 Mar 24. PMID 23996808
- [Background] Koo BK, Kim D, Joo SK, Kim JH, Chang MS, Kim BG, Lee KL, Kim W. Sarcopenia is an independent risk factor for non-alcoholic steatohepatitis and significant fibrosis. J Hepatol. 2017 Jan;66(1):123-131. doi: 10.1016/j.jhep.2016.08.019. Epub 2016 Sep 4. PMID 27599824
- [Background] Kim G, Lee SE, Lee YB, Jun JE, Ahn J, Bae JC, Jin SM, Hur KY, Jee JH, Lee MK, Kim JH. Relationship Between Relative Skeletal Muscle Mass and Nonalcoholic Fatty Liver Disease: A 7-Year Longitudinal Study. Hepatology. 2018 Nov;68(5):1755-1768. doi: 10.1002/hep.30049. Epub 2018 Oct 14. PMID 29679374
- [Background] Lee MJ, Kim EH, Bae SJ, Kim GA, Park SW, Choe J, Jung CH, Lee WJ, Kim HK. Age-Related Decrease in Skeletal Muscle Mass Is an Independent Risk Factor for Incident Nonalcoholic Fatty Liver Disease: A 10-Year Retrospective Cohort Study. Gut Liver. 2019 Jan 15;13(1):67-76. doi: 10.5009/gnl18070. PMID 30037166
- [Background] Cai C, Song X, Chen Y, Chen X, Yu C. Relationship between relative skeletal muscle mass and nonalcoholic fatty liver disease: a systematic review and meta-analysis. Hepatol Int. 2020 Jan;14(1):115-126. doi: 10.1007/s12072-019-09964-1. Epub 2019 Jul 9. PMID 31290072
- [Background] De Fre CH, De Fre MA, Kwanten WJ, Op de Beeck BJ, Van Gaal LF, Francque SM. Sarcopenia in patients with non-alcoholic fatty liver disease: is it a clinically significant entity? Obes Rev. 2019 Feb;20(2):353-363. doi: 10.1111/obr.12776. Epub 2018 Nov 25. PMID 30474288
- [Background] Pacifico L, Perla FM, Chiesa C. Sarcopenia and nonalcoholic fatty liver disease: a causal relationship. Hepatobiliary Surg Nutr. 2019 Apr;8(2):144-147. doi: 10.21037/hbsn.2018.11.11. No abstract available. PMID 31098363
- [Background] Bhanji RA, Narayanan P, Allen AM, Malhi H, Watt KD. Sarcopenia in hiding: The risk and consequence of underestimating muscle dysfunction in nonalcoholic steatohepatitis. Hepatology. 2017 Dec;66(6):2055-2065. doi: 10.1002/hep.29420. Epub 2017 Oct 30. PMID 28777879
- [Background] Pelusi S, Valenti L. Building mass to prevent non-alcoholic fatty liver disease? Hepatobiliary Surg Nutr. 2019 Apr;8(2):173-176. doi: 10.21037/hbsn.2018.12.07. No abstract available. PMID 31098372
- [Background] Hardee JP, Lynch GS. Current pharmacotherapies for sarcopenia. Expert Opin Pharmacother. 2019 Sep;20(13):1645-1657. doi: 10.1080/14656566.2019.1622093. Epub 2019 May 23. PMID 31120352
- [Background] Nachit M, Leclercq IA. Emerging awareness on the importance of skeletal muscle in liver diseases: time to dig deeper into mechanisms! Clin Sci (Lond). 2019 Feb 12;133(3):465-481. doi: 10.1042/CS20180421. Print 2019 Feb 14. PMID 30755499
- [Background] Cabrera D, Cabello-Verrugio C, Solis N, San Martin D, Cofre C, Pizarro M, Arab JP, Abrigo J, Campos F, Irigoyen B, Carrasco-Avino G, Bezares K, Riquelme V, Riquelme A, Arrese M, Barrera F. Somatotropic Axis Dysfunction in Non-Alcoholic Fatty Liver Disease: Beneficial Hepatic and Systemic Effects of Hormone Supplementation. Int J Mol Sci. 2018 May 2;19(5):1339. doi: 10.3390/ijms19051339. PMID 29724029
- [Background] Wong VW, Adams LA, de Ledinghen V, Wong GL, Sookoian S. Noninvasive biomarkers in NAFLD and NASH - current progress and future promise. Nat Rev Gastroenterol Hepatol. 2018 Aug;15(8):461-478. doi: 10.1038/s41575-018-0014-9. PMID 29844588
- [Background] Ruffillo G, Fassio E, Alvarez E, Landeira G, Longo C, Dominguez N, Gualano G. Comparison of NAFLD fibrosis score and BARD score in predicting fibrosis in nonalcoholic fatty liver disease. J Hepatol. 2011 Jan;54(1):160-3. doi: 10.1016/j.jhep.2010.06.028. Epub 2010 Aug 22. PMID 20934232
- [Background] Perez-Gutierrez OZ, Hernandez-Rocha C, Candia-Balboa RA, Arrese MA, Benitez C, Brizuela-Alcantara DC, Mendez-Sanchez N, Uribe M, Chavez-Tapia NC. Validation study of systems for noninvasive diagnosis of fibrosis in nonalcoholic fatty liver disease in Latin population. Ann Hepatol. 2013 May-Jun;12(3):416-24. PMID 23619258
- [Background] Goulart AC, Oliveira IR, Alencar AP, Santos MS, Santos IS, Martines BM, Meireles DP, Martines JA, Misciagna G, Bensenor IM, Lotufo PA. Diagnostic accuracy of a noninvasive hepatic ultrasound score for non-alcoholic fatty liver disease (NAFLD) in the Brazilian Longitudinal Study of Adult Health (ELSA-Brasil). Sao Paulo Med J. 2015 Mar-Apr;133(2):115-24. doi: 10.1590/1516-3180.2014.9150812. Epub 2015 Apr 1. PMID 26018881
- [Background] Perazzo H, Bensenor I, Mill JG, Pacheco AG, da Fonseca MJM, Griep RH, Lotufo P, Chor D. Prediction of Liver Steatosis Applying a New Score in Subjects from the Brazilian Longitudinal Study of Adult Health. J Clin Gastroenterol. 2020 Jan;54(1):e1-e10. doi: 10.1097/MCG.0000000000001007. PMID 29505553
- [Background] Tovo CV, Villela-Nogueira CA, Leite NC, Panke CL, Port GZ, Fernandes S, Buss C, Coral GP, Cardoso AC, Cravo CM, Calcado FL, Rezende GFM, Ferreira FC, Araujo-Neto JM, Perez RM, Moraes-Coelho HS, de Mattos AA. Transient hepatic elastography has the best performance to evaluate liver fibrosis in non-alcoholic fatty liver disease (NAFLD). Ann Hepatol. 2019 May-Jun;18(3):445-449. doi: 10.1016/j.aohep.2018.09.003. Epub 2019 Apr 12. PMID 31031166
- [Background] Yilmaz Y, Ergelen R, Akin H, Imeryuz N. Noninvasive detection of hepatic steatosis in patients without ultrasonographic evidence of fatty liver using the controlled attenuation parameter evaluated with transient elastography. Eur J Gastroenterol Hepatol. 2013 Nov;25(11):1330-4. doi: 10.1097/MEG.0b013e3283623a16. PMID 23660937
- [Background] Zhang X, Wong GL, Wong VW. Application of transient elastography in nonalcoholic fatty liver disease. Clin Mol Hepatol. 2020 Apr;26(2):128-141. doi: 10.3350/cmh.2019.0001n. Epub 2019 Nov 8. PMID 31696690
- [Background] Benedict M, Zhang X. Non-alcoholic fatty liver disease: An expanded review. World J Hepatol. 2017 Jun 8;9(16):715-732. doi: 10.4254/wjh.v9.i16.715. PMID 28652891
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. J Hepatol. 2016 Jun;64(6):1388-402. doi: 10.1016/j.jhep.2015.11.004. Epub 2016 Apr 7. No abstract available. PMID 27062661
- [Background] Wong VW, Chan WK, Chitturi S, Chawla Y, Dan YY, Duseja A, Fan J, Goh KL, Hamaguchi M, Hashimoto E, Kim SU, Lesmana LA, Lin YC, Liu CJ, Ni YH, Sollano J, Wong SK, Wong GL, Chan HL, Farrell G. Asia-Pacific Working Party on Non-alcoholic Fatty Liver Disease guidelines 2017-Part 1: Definition, risk factors and assessment. J Gastroenterol Hepatol. 2018 Jan;33(1):70-85. doi: 10.1111/jgh.13857. No abstract available. PMID 28670712
- [Background] Cabezas J, Bataller R. Alcoholic liver disease: New UK alcohol guidelines and Dry January: enough to give up boozing? Nat Rev Gastroenterol Hepatol. 2016 Apr;13(4):191-2. doi: 10.1038/nrgastro.2016.39. Epub 2016 Mar 9. No abstract available. PMID 26956065
- [Background] Crabb DW, Im GY, Szabo G, Mellinger JL, Lucey MR. Diagnosis and Treatment of Alcohol-Associated Liver Diseases: 2019 Practice Guidance From the American Association for the Study of Liver Diseases. Hepatology. 2020 Jan;71(1):306-333. doi: 10.1002/hep.30866. No abstract available. PMID 31314133
- [Background] Dash A, Figler RA, Sanyal AJ, Wamhoff BR. Drug-induced steatohepatitis. Expert Opin Drug Metab Toxicol. 2017 Feb;13(2):193-204. doi: 10.1080/17425255.2017.1246534. Epub 2016 Oct 27. PMID 27759439
- [Background] Davis R, Campbell R, Hildon Z, Hobbs L, Michie S. Theories of behaviour and behaviour change across the social and behavioural sciences: a scoping review. Health Psychol Rev. 2015;9(3):323-44. doi: 10.1080/17437199.2014.941722. Epub 2014 Aug 8. PMID 25104107
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] Anderson ES, Winett RA, Wojcik JR. Self-regulation, self-efficacy, outcome expectations, and social support: social cognitive theory and nutrition behavior. Ann Behav Med. 2007 Nov-Dec;34(3):304-12. doi: 10.1007/BF02874555. PMID 18020940
- [Background] Nagpal TS, Prapavessis H, Campbell C, Mottola MF. Measuring Adherence to a Nutrition and Exercise Lifestyle Intervention: Is Program Adherence Related to Excessive Gestational Weight Gain? Behav Anal Pract. 2017 May 17;10(4):347-354. doi: 10.1007/s40617-017-0189-5. eCollection 2017 Dec. PMID 29214130
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Ryan MC, Itsiopoulos C, Thodis T, Ward G, Trost N, Hofferberth S, O'Dea K, Desmond PV, Johnson NA, Wilson AM. The Mediterranean diet improves hepatic steatosis and insulin sensitivity in individuals with non-alcoholic fatty liver disease. J Hepatol. 2013 Jul;59(1):138-43. doi: 10.1016/j.jhep.2013.02.012. Epub 2013 Feb 26. PMID 23485520
- [Background] Thoma C, Day CP, Trenell MI. Lifestyle interventions for the treatment of non-alcoholic fatty liver disease in adults: a systematic review. J Hepatol. 2012 Jan;56(1):255-66. doi: 10.1016/j.jhep.2011.06.010. Epub 2011 Jul 1. PMID 21723839